CLINICAL TRIAL: NCT01580800
Title: National Breast Cancer and Lymphedema Registry
Status: Terminated | Type: Observational
Why Stopped: Low enrollment, incomplete participant data, and follow-up information
Sponsor: Stanley Rockson (Other)
Responsible Party: Sponsor-Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: SU-10042011-8529; 22349 (Other: Stanford University)
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer survivors: Patients who have undergone breast cancer treatment (e.g. surgery, node dissection, chemotherapy and/or radiation therapy), and what affect this has had on their arm health.

SUMMARY:
The purpose of the National Breast Cancer Lymphedema Registry is to collect health information in order to study the lymphedema as a complication of breast cancer treatment. The investigators hope to learn whether early diagnosis will help to prevent lymphedema or, if it does occur, to reduce the severity.

DETAILED DESCRIPTION:
Historically, breast cancer-associated lymphedema has been relatively ignored, with mis-diagnosis, late diagnosis, and failure to treat. The condition has a measurable, substantial impact on patient function and perceived quality of life (QOL). Recent pilot studies suggest that interventions that are designed to facilitate early diagnosis and preventive strategies have a major impact on the incidence and severity of disease burden. This registry is designed to prospectively capture the relevant data to document the impact of preemptive diagnostic and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivorship

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Preemptive diagnostic and treatment strategies | Each enrolled patient will be followed for an average of 1 year
  The methods for lymphedema surveillance and detection will be correlated to the new appearance of lymphedema in this cohort of breast cancer survivors. We will also assess severity of lymphedema and responsiveness to treatment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Stanford Healthcare Lymphedema Clinic — http://stanfordhealthcare.org/medical-conditions/blood-heart-circulation/lymphedema.html